CLINICAL TRIAL: NCT01992549
Title: Extension Study for Patients Who Completed GENA-05 (NuProtect)- to Investigate Immunogenicity, Efficacy and Safety of Treatment With Human-cl rhFVIII
Brief Title: Study to Investigate Immunogenicity, Efficacy and Safety of Treatment With Human-cl rhFVIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENA-15
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Severe Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human-cl rhFVIII (Experimental)
  Interventions: Biological: Human-cl rhFVIII

INTERVENTIONS:
Biological: Human-cl rhFVIII

SUMMARY:
The purpose of the study is to collect long-term data on the inhibitor development rate of Human-cl rhFVIII in previously untreated patients with severe Hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who completed GENA-05 in accordance with the study protocol

Exclusion Criteria:

1. Severe liver or kidney disease
2. Concomitant treatment with any systemic immunosuppressive drug;
3. Other FVIII concentrate than Human-cl rhFVIII was received between completion visit of GENA-05 and start of GENA-15 (except emergency cases).

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-04; Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sigurd Knaub, PhD, Study Director — Octapharma
Locations (15):
- UC Davis Medical Center, Sacramento, California, United States
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Hospital for Sick Children, Toronto
- France (2):
  - Hopital de la Timone, Marseille
  - Hôpital Kremlin Bicètre, Paris
- Institute of Hematology and Transfusiology, Tbilisi, Georgia
- India (2):
  - Sahyadri Speciality Hospital, Pune
  - Christian Medical College, Vellore
- IMSP Mother and Child Institute, Chisinau, Moldova
- University Medical School, Warsaw, Poland
- Ukraine (2):
  - The National Children Specialized Hospital "OHMATDET", Kiev
  - Danylo Halytsky Lviv National Medical University, Lviv
- Great Ormond Street Hospital for Children, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Human-cl rhFVIII: Of the total number of patients that started in the study, all those in the safety (SAF) population received at least 1 infusion of Human-cl rhFVIII. Patients who had data collected post-treatment were included in the intent-to-treat (ITT) population. Prophylactic treatment dose given to all patients in the PROPH population (all patients who received at least 1 administration of Human-cl rhFVIII with prophylaxis documented as the reason for treatment): >20 IU FVIII/kg body weight (BW). On-demand treatment of bleeding episodes (BEs) dose given to the BLEED population (all patients with bleeding episodes treated with Human-cl rhFVIII): 20-30 IU FVIII/kg BW (minor haemorrhage), 30-40 IU FVIII/kg BW (moderate to major haemorrhage) or 50-80 IU FVIII/kg BW (major to life-threatening haemorrhage). Surgical prophylaxis dose was given to the SURG population (all patients with surgeries treated with Human-cl rhFVIII): 25-30 IU FVIII/kg BW (minor surgeries); >50 IU FVIII/kg BW (major surgeries).
Period: Overall Study
Arm/Group | Human-cl rhFVIII
Started | 48
SAF Population (SAF population = study population of patients in safety analysis) | 48
ITT Population (ITT population = intent-to-treat population) | 47
PROPH Population (PROPH population = study population of patients receiving prophylaxis) | 47
BLEED Population (BLEED population = study population of Bleeding Events (BEs)) | 29
SURG Population (SURG population = study population of patients undergoing surgery treated with Human-cl rhFVIII) | 3
Completed | 44
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Serious Adverse Event | 1
Not completed — Product Switch to Extend Half Life | 1

BASELINE CHARACTERISTICS:
Population: The safety (SAF) population consist of all patients who received at least one infusion of Human-cl rhFVIII (n=48).
Groups:
- Human-cl rhFVIII: The safety (SAF) population consist of all patients who received at least one infusion of Human-cl rhFVIII (n=48).
Arm/Group | Human-cl rhFVIII
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.47 (2.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 2
  Unknown or Not Reported | 0
Body Mass Index (BMI) at screening [Mean (Full Range); unit: kg/m^2] | 16.46 [12.4 to 22.3]
Height at screening [Mean (Full Range); unit: Centimeters (cm)] | 97.44 [78 to 138]
Weight at screening [Mean (Full Range); unit: Kilograms (kg)] | 15.84 [9.1 to 33.0]
Family history of inhibitors [Count of Participants; unit: Participants]
  Yes | 3
  No | 45

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity of Human-cl rhFVIII: Incidence of Inhibitors
Description: The number of patients developing FVIII inhibitors was observed during the observation period by assessing inhibitor development by the modified Bethesda assay (Nijmegen modification) using congenital FVIII-deficient human plasma spiked with Human-cl rhFVIII. The definition threshold for a "positive" inhibitor was if the modified Bethesda assay resulted in a titre ≥0.6 BU/mL at any time point during the observation period.
Time Frame: Maximum two years
Population: The analysis was performed for the safety (SAF) population which includes all patients who received at least 1 infusion of Human-cl rhFVIII (N=48)
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Human-cl rhFVIII: The safety (SAF) population consist of all patients who received at least one infusion of Human-cl rhFVIII
Arm/Group | Human-cl rhFVIII
Number analyzed (Participants) | 48
participants | 0 [0.000 to 7.549]

2. Secondary Outcome: Frequency of Spontaneous Break-through Bleeds
Description: The annualized bleeding rate (ABR) was calculated during the time of prophylactic treatment with Human-cl rhFVIII for spontaneous bleeding events (BEs).
Time Frame: Maximum 2 years
Population: The analysis population includes all patients in PROPH population who received at least one prophylactic treatment with Human-cl rhFVIII (n=47).
Measure: Mean (95% Confidence Interval); unit: Events/year (ABR)
Groups:
- ITT/PROPH Population: All patients who had data collected post-treatment with Human-cl rhFVIII and at least one prophylactic treatment with Human-cl rhFVIII (n=47).
Arm/Group | ITT/PROPH Population
Number analyzed (Participants) | 47
Events/year (ABR) | 0.283 [0.153 to 0.527]

3. Secondary Outcome: Efficacy of Human-cl rhFVIII for the Treatment of Bleeds
Description: A personal efficacy assessment (final outcome) to assess the efficacy of Human-cl rhFVIII for the on-demand treatment of bleeding episodes (BEs) at the end of a BE. Efficacy was assessed using a four-point scale (excellent, good, moderate, none) by the patient's parent(s)/legal guardian(s) together with the investigator in case of on site treatment.
Time Frame: Maximum 2 years
Population: The analysis population included all patients who received on-demand treatment with Human-cl rhFVIII for bleeding episodes (BLEED population; n=29).
Measure: Count of Units; unit: Bleeding episodes
Units Other Than Participants: Bleeding episodes
Groups:
- BLEED Population: All patients that experienced at least one bleeding episode treated with Human-cl rhFVIII (n=29)
Arm/Group | BLEED Population
Number analyzed (Participants) | 29
Number analyzed (Bleeding episodes) | 111
Bleeding episodes
  Excellent | 58
  Good | 28
  Moderate | 21
  None | 3
  Not done | 1

4. Secondary Outcome: Efficacy of Human-cl rhFVIII for Surgical Prophylaxis
Description: An overall efficacy assessment to assess the efficacy of human-cl rhFVIII in surgical prophylaxis of minor and major surgeries. The efficacy assessment was analyzed using a four-point scale (excellent, good, moderate, none). If surgeries could not be assessed due to limited data available or having taken place outside the study site, the results were classified as "not done".
Time Frame: Maximum 2 years
Population: The analysis population includes 3 patients that received Human-cl rhFVIII for surgical prophylaxis during a total of 4 surgeries (SURG population). Of these, 1 patient had two minor surgeries and 2 patients had one major surgery each.
Measure: Count of Units; unit: Surgeries
Units Other Than Participants: Surgeries
Groups:
- Minor Surgeries: All patients that had minor surgeries performed under Human-cl rhFVIII treatment (n=1)
- Major Surgeries: All patients that had major surgeries performed under Human-cl rhFVIII treatment (n=2)
- SURG Population: All patients that had surgeries performed under Human-cl rhFVIII treatment (n=3)
Arm/Group | Minor Surgeries | Major Surgeries | SURG Population
Number analyzed (Participants) | 1 | 2 | 3
Number analyzed (Surgeries) | 2 | 2 | 4
Surgeries
  Excellent | 0 | 2 | 2
  Good | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  None | 0 | 0 | 0
  Not done | 2 | 0 | 2

5. Secondary Outcome: The Occurrence of Any Adverse Event (AE)
Description: The frequency of AEs, as monitored throughout the whole study by the number of patients with at least one adverse event occurrence.
Time Frame: Maximum 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- SAF Population: The safety (SAF) population consist of all patients who received at least one infusion of Human-cl rhFVIII (n=48).
Arm/Group | SAF Population
Number analyzed (Participants) | 48
Participants
  Adverse event | 29
  Serious adverse event (SAE) | 5
  Severe AE | 3
  Temporally related adverse event | 20
  Death | 0
  AE leading to permanent discontinuation | 1

ADVERSE EVENTS:
Time Frame: Maximum 2 years
Arm/Group | SAF Population
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 5/48
Other Adverse Events (participants affected / at risk) | 29/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAF Population (N=48)
Pneumonia (Infections and infestations) | 2
Varicella (Infections and infestations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage (Vascular disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.08% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAF Population (N=48)
Nasopharyngitis (Infections and infestations) | 10
Varicella (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 4
Ear infection (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 4
Tonsillitis (Infections and infestations) | 3
Otitis media (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Pulpitis dental (Infections and infestations) | 2
Respiratory tract infection viral (Infections and infestations) | 2
Tracheitis (Infections and infestations) | 2
Pyrexia (General disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Octapharma agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Octapharma supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial. Octapharma also reserves the right to review data prior to publishing and provide comments/changes within a certain time period.

DOCUMENTS (2):
  • Study Protocol (2013-09-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT01992549/Prot_002.pdf
  • Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT01992549/SAP_003.pdf